CLINICAL TRIAL: NCT01700842
Title: Multicenter Study of Antimicrobial Resistance of Gram-positive and Gram-negative Clinical Strains to Ceftaroline and Other Antimicrobials in Russia
Acronym: CERBERUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-IRU-XXX-2012/1
Record Dates: First submitted 2012-10-03; First posted 2012-10-04 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Bacterial Skin Diseases
Keywords: ceftaroline, infection, CAPB, CAP, ABSSSI, cSSTI
MeSH Terms: conditions — Skin Diseases, Bacterial; Infections

STUDY DESIGN:
Biospecimen Retention: None Retained — Microbiological strains

SUMMARY:
Approximately 3,000 of clinically significant isolates of different species from respective respective sources in geographically distinct Russian cities will be collected and tested on ceftaroline and other antimicrobials.

ELIGIBILITY:
Inclusion Criteria:

* Isolates derived from patients' clinical material will be included in the study
* Isolates collected retro- and prospectively will be included in the study (from 01.01.2008 till 31.12.2012)
* Isolates, allocated of a clinical material of adult patients (> 18 years), should make not less than 70 % from total number of included isolates)
* All included isolates should be unique: only one isolate can be included in the study of each biological type from each patient
* All isolates should correspond to clinic-laboratory criteria of the etiologic importance, i.e. should be derived from patients with infection symptoms from the corresponding clinical material
* Case report form (CRF) (Appendix 1) should be correctly completed for each isolate

Exclusion Criteria:

* ESBL-producing representatives of Enterobacteriaceae (ESBL-Extended-spectrum beta-lactamase)
* Isolates, arrived in the central laboratory contaminated or unviable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: clinical material form patients in geographically distinct Russian cities
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage(numerical) MIC distribution of microorganisms for ceftaroline and other tested antimicrobials, including MIC50 and MIC90, percent(quantity)of susceptible and resistant strains in accordance with EUCAST or CLSI recommended breakpoints. | up to 3 months
  MIC- Minimum inhibitory concentration; EUCAST - European Committee on Antimicrobial Susceptibility Testing; CLSI- Clinical and Laboratory Standard Institute

SECONDARY OUTCOMES:
Percentage(numerical)MIC distribution of microorganisms,including MIC50 and MIC90, percent(quantity) of susceptible and resistant strains, to tested antibiotics depend on: infection localization, medical condition, ward/unit profile,patient profile(age) | up to 3 months
Percentage(numerical)MIC distribution of microorganisms,including MIC50 and MIC90, percent(quantity) of susceptible and resistant strains,to ceftaroline and other antimicrobials by years from 2008 to 2012 | upto 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Research Site, Saint Petersburg
  - Research Site, Smolensk